CLINICAL TRIAL: NCT03310216
Title: The Clinical Application of Artificial Intelligent Visual Inspection System
Brief Title: The Clinical Application of Artificial Intelligent(AI) Visual Inspection System
Acronym: AI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CCPMOH2017-China-8
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Ophthalmology
Keywords: artificial intelligent; visual inspection

STUDY DESIGN:
Intervention Model Description: Patients are assigned to two groups: participants in group I are provided AI visual inspection system first and EDTRS later, while in Group II, the participants are provided EDTRS first and AI visual inspection system later.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order I of visual inspection (Experimental): Participants in group I are provided AI visual inspection system first and EDTRS later.
  Interventions: Procedure: Order I of visual inspection
- Order II of visual inspection (Active Comparator): Participants in group II are provided EDTRS first and AI visual inspection system later.
  Interventions: Procedure: Order II of visual inspection

INTERVENTIONS:
Procedure: Order I of visual inspection — Participants in group I are provided AI visual inspection system first and EDTRS later.
  Arms: Order I of visual inspection
Procedure: Order II of visual inspection — The participants in Group II are provided EDTRS first and AI visual inspection system later.
  Arms: Order II of visual inspection

SUMMARY:
In this study, the investigators provide participants from ophthalmic clinic the AI visual inspection system and EDTRS in the purpose of seeking out a better way of visual inspection with high efficiency and accuracy, and report a prospective, randomized controlled study aiming at comparison of AI visual inspection system and EDTRS for visual inspection.

DETAILED DESCRIPTION:
Patients ≤90 years old from ophthalmic clinic are enrolled to a prospective, randomized controlled study. Patients are assigned to two groups: participants in group I are provided AI visual inspection system first and EDTRS later, while in Group II, the participants are provided EDTRS first and AI visual inspection system later. All of the visual inspection methods will be repeated two times. Investigators compare the accuracy and repeatability of the AI visual inspection system, time consuming, costs and the satisfaction level between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients≤90 years old from ophthalmic clinic; Written informed consents provided

Exclusion Criteria:

* Can not cooperate with the visual inspection; Unwilling to participate in this trail

Ages: 1 Month to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The accuracy of AI visual inspection system | Baseline
  The accuracy of AI visual inspection system was calculated.

SECONDARY OUTCOMES:
The time taken of visual inspection | Baseline
  The time taken of visual inspection was calculated.
Costs of AI visual inspection system | Baseline
  Costs of AI visual inspection system was calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China